CLINICAL TRIAL: NCT04642417
Title: Effectiveness of Experiential Learning on Dietary Fiber Literacy and Bowel Symptom Management After Surgery for Colorectal Cancer
Brief Title: Effectiveness of Experiential Learning on Dietary Fiber Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202008045RINC
Record Dates: First submitted 2020-11-05; First posted 2020-11-24 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2021-12

CONDITIONS: Literacy; Bowel Symptoms
Keywords: Colorectal cancer surgery; Literacy; Dietary fiber food literacy; Dietary fiber; experiential learning
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned (1:1) to routine or EL group. EL group received simulated dietary-fiber experiential learning and one dietary application consultation session one month post-surgery, in addition to routine care before discharge.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Using a randomization design, investigators randomly placed the number into the envelope. This procedure was concealed from the provider or patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): intervention give experience dietary fiber literacy
  Interventions: Other: dietary fiber literacy; Other: routine care
- No Intervention (No Intervention): give standard education

INTERVENTIONS:
Other: dietary fiber literacy — education
  Arms: Experimental
Other: routine care — routine care
  Arms: Experimental

SUMMARY:
Acute symptom onset is the most common problem in colorectal cancer surgery, and it is also the source of the most painful impact on patients' lives. The second is the fear of cancer recurrence and complications, and psychological problems such as fear or depression are prone to occur. Studies have found that colorectal cancer is gradually suffering from complications and symptoms for six months, and even uncontrollable gas, leakage and incontinence, causing frequent occurrence of underwear. , The body and mind are severely impacted, and affect daily activities and quality of life. The problem of initial symptom management after colorectal cancer surgery is highly complex, and patients even have to self-manage diseases and symptoms in the face of physical and psychological adjustment. The provision and consultation of knowledge and information from nursing staff can prepare patients for discharge and meet their needs for knowledge and information, and can help patients achieve effective self-management capabilities.The foundation of health awareness emphasizes health knowledge. Health awareness is a more advanced knowledge achievement; it is the ability to make judgments and decisions in daily life related to health care, disease prevention and health promotion, and is the basic element of achieving self-management of health. Dietary knowledge is also a higher-level knowledge, which reflects dietary knowledge in behavior, food choices and criticism, and reflects on food choices and health decisions. Insufficient dietary knowledge will affect food choices, judgments and decisions, resulting in insufficient diet-related knowledge.Studies have confirmed that the health-related knowledge of cancer patients is significantly related to disease self-management. Only when patients understand their own diseases can they actively participate in self-health management. Nursing staff play a pivotal role in the care of patients with colorectal cancer. Through the knowledge transfer of nursing staff and guiding patients to take care of themselves, they can help improve postoperative dietary intake behaviors, thereby enhancing dietary awareness. Literature review of chronic disease self-management, nursing staff provide patients with sufficient relevant knowledge education, which can enhance patients' self-efficacy and enhance disease self-management ability.

DETAILED DESCRIPTION:
Through the re-giving and encouragement of knowledge information, personal behavior control and reframing can be achieved, which can be effective To promote personal health. Nursing staff's consultation and face-to-face interviews can significantly improve patients' health-related knowledge, effective education strategies and assist patients in self-management of disease-related problems.

Experiential learning interaction can deepen the patient's impression and memory, improve the patient's knowledge and skills about the disease, increase patient participation in self-decision-making, improve self-efficacy, present better health-related knowledge, and achieve self-management capabilities. Past studies have also found that telephone tracking and consultation, emails, and giving diet manuals can help patients with colorectal cancer make significant changes in their healthy diet choices.

ELIGIBILITY:
inclusion criteria

1. You can read the newspaper yourself.
2. Emotions and cognitive functions can be answered without barriers
3. After clinical diagnosis of colorectal cancer (stage I-III), the doctor has recommended and arranged for colorectal cancer Surgery.
4. Age between 20 to 85 years old.
5. Willing to use a computer tablet to conduct a questionnaire survey.

exclusion criteria

1. Those who are currently receiving chemical drugs or radiation therapy.
2. Clinical diagnosis of colorectal cancer stage IV (stage IV); recurrence, metastasis or other cancers
3. Diagnosis of mental illness patients.
4. Cannot read the newspaper on their own

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Bowel Symptom | 20 minutes
  LARS; minimum to maximum scores by 5-42, higher is mean severe bowel symptoms

SECONDARY OUTCOMES:
Dietary Fiber food Literacy | 50 minutes
  Dietary Fiber Literacy scale；the maximum scores is 41, higher is better
food frequency | 20 minutes
  food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Been-Ren Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan